CLINICAL TRIAL: NCT00391053
Title: Phase III Lot Consistency, Immunogenicity and Safety Study of Three Lots of Fluzone High Dose Vaccine Compared With One Lot of Standard Fluzone® in Adults ≥ 65 Years of Age.
Brief Title: Immunogenicity of High-dose Inactivated, Split-virion Influenza Vaccine Versus Standard Fluzone Vaccine in the Elderly
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: FIM05
Record Dates: First submitted 2006-10-20; First posted 2006-10-23 (Estimated); Results first posted 2010-04-30 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2016-04

CONDITIONS: Orthomyxoviridae Infection; Influenza; Myxovirus Infection
Keywords: Influenza; Orthomyxoviruses; Inactivated Split-virion influenza vaccine; Adults
MeSH Terms: conditions — Orthomyxoviridae Infections; Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Study Group 1 (Experimental): Participants will receive the High-Dose Inactivated, Split-Virion Influenza Vaccine Lot 1
  Interventions: Biological: High-Dose Inactivated, Split-Virion Influenza Vaccine
- Study Group 2 (Experimental): Participants will receive the High-Dose Inactivated, Split-Virion Influenza Vaccine Lot 2
  Interventions: Biological: High-Dose Inactivated, Split-Virion Influenza Vaccine
- Study Group 3 (Experimental): Participants will receive the High-Dose Inactivated, Split-Virion Influenza Vaccine Lot 3
  Interventions: Biological: High-Dose Inactivated, Split-Virion Influenza Vaccine
- Group 4 (Active Comparator): Participants will receive the Standard Fluzone® vaccine
  Interventions: Biological: Inactivated, Split-Virion Influenza Vaccine

INTERVENTIONS:
Biological: High-Dose Inactivated, Split-Virion Influenza Vaccine — 0.5 mL, IM
  Other Names: Fluzone® High-Dose
  Arms: Study Group 1
Biological: High-Dose Inactivated, Split-Virion Influenza Vaccine — 0.5 mL, IM
  Other Names: Fluzone® High-Dose
  Arms: Study Group 2
Biological: High-Dose Inactivated, Split-Virion Influenza Vaccine — 0.5 mL, IM
  Other Names: Fluzone® High-Dose
  Arms: Study Group 3
Biological: Inactivated, Split-Virion Influenza Vaccine — 0.5 mL, IM
  Other Names: Fluzone® 2006-2007 formulation
  Arms: Group 4

SUMMARY:
Compared to young adults, the elderly mount a lower antibody response to vaccination. Thus, improvement of the immune response to influenza vaccination in this age group, which is at higher risk for influenza-related morbidity and mortality, represents an important unmet need.

Primary Objectives:

Immunogenicity:

* To demonstrate lot consistency of the Fluzone High Dose (Fluzone HD) manufacturing process through evaluation of the immune responses elicited by three different lots.
* To demonstrate the superiority of Fluzone HD vaccine compared to standard-dose Fluzone® vaccine.

Secondary Objectives:

Immunogenicity:

* To describe the seroprotection of Fluzone HD compared to that of standard dose Fluzone® vaccine.

Safety:

* To describe the safety profile of Fluzone HD, in terms of solicited -, unsolicited adverse and serious adverse events post-vaccination.
* To describe clinical information on some additional defined criteria during the six months following vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 65 years on the day of vaccination.
* Informed consent form signed.
* Medically stable. (Subjects may have underlying chronic conditions such as hypertension, diabetes, ischemic heart disease, or hypothyroidism, as long as their symptoms/signs are controlled. If they are on medication for a condition, the medication dose must have been stable for at least 3 weeks preceding vaccination.)
* Able to attend all scheduled visits and to comply with all trial procedures.

Exclusion Criteria:

* Systemic hypersensitivity to eggs, chicken proteins, or any of the vaccine components, or a history of a life-threatening reaction to the standard-dose Fluzone® vaccine or a vaccine containing any of the same substances.
* Congenital or history of acquired immunodeficiency, or immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within the preceding six months.
* Systemic corticosteroid therapy, as follows:

Continuous use with a dosage equivalent to > 15 mg/day of oral prednisone for 90 days preceding vaccination.

Sporadic use with a dosage equivalent to > 40 mg/day of oral prednisone for > 14 consecutive days in the 90 days preceding vaccination.

Note:Use of topical or inhalant corticosteroids is acceptable.

* Neoplastic disease or any hematologic malignancy (except localized skin or prostate cancer that is stable at the time of vaccination in the absence of therapy, as well as subjects who have a history of neoplastic disease and who have been disease-free for ≥ 5 years).
* Current alcohol abuse or drug addiction that in the opinion of the investigator may interfere with the subject's ability to comply with trial procedures.
* Receipt of blood or blood-derived products in the past three months.
* Participation in a trial of a high-dose influenza vaccine in the past 12 months.
* Receipt of influenza vaccine in the past six months.
* Receipt of any other vaccine in the past four weeks.
* Planned receipt of any other vaccine in the four weeks following the trial vaccination.
* Participation in another clinical trial in the past four weeks.
* Planned participation in another clinical trial during the present trial period.

Note:Concomitant participation in an observational trial (not involving drugs, vaccines, or medical devices) is acceptable.

* Thrombocytopenia or bleeding disorder contraindicating intramuscular (IM) vaccination.
* History of Guillain-Barré syndrome.
* Subject deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized without his/her consent.
* An acute febrile illness (oral temperature ≥ 99.5ºF [≥ 37.5ºC]) within 24 hours prior to vaccination. If this contraindication exists, vaccination will be deferred until the participant has been afebrile for at least 24 hours.
* Signs and symptoms of an acute infectious respiratory illness. If this exists, vaccination will be deferred until the symptoms resolve.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 3851 (Actual)
Dates: Start 2006-10; Primary Completion 2007-07 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Inc.
Locations (28):
- United States (28):
  - Mesa, Arizona
  - Phoenix, Arizona
  - Tempe, Arizona
  - Tucson, Arizona
  - San Diego, California
  - Stratford, Connecticut
  - Clearwater, Florida
  - Coral Gables, Florida
  - Orlando, Florida
  - Pembroke Pines, Florida
  - Wichita, Kansas
  - Rockville, Maryland
  - Rochester, Minnesota
  - Kansas City, Missouri
  - St Louis, Missouri
  - Endwell, New York
  - Rochester, New York
  - Cary, North Carolina
  - Raleigh, North Carolina
  - Downington, Pennsylvania
  - Erie, Pennsylvania
  - Warwick, Rhode Island
  - Dallas, Texas
  - Plano, Texas
  - West Jordan, Utah
  - Norfolk, Virginia
  - Richmond, Virginia
  - Marshfield, Wisconsin

REFERENCES:
- [Result] Falsey AR, Treanor JJ, Tornieporth N, Capellan J, Gorse GJ. Randomized, double-blind controlled phase 3 trial comparing the immunogenicity of high-dose and standard-dose influenza vaccine in adults 65 years of age and older. J Infect Dis. 2009 Jul 15;200(2):172-80. doi: 10.1086/599790. PMID 19508159
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from 09 October 2006 to 21 December 2006 at 30 US sites.
Pre-assignment Details: A total of 3851 participants who met the inclusion and exclusion criteria were randomized and vaccinated. The vaccine received by 14 participants could not be verified, they were excluded from all analyses except immunogenicity analysis. 4 participants that started the study, but had no post-vaccination assessment were also excluded from analysis.
Groups:
- High-Dose Inactivated, Split-Virion Influenza Vaccine Lot 1: Participants aged 65 years or older at enrollment, treated with high-dose trivalent inactivated influenza vaccine (Fluzone HD) 2006-2007 formulation, Lot 1
- High-Dose Inactivated, Split-Virion Influenza Vaccine Lot 2: Participants aged 65 years or older at enrollment, treated with high-dose trivalent inactivated influenza vaccine (Fluzone HD) 2006-2007 formulation, Lot 2
- High-Dose Inactivated, Split-Virion Influenza Vaccine Lot 3: Participants aged 65 years or older at enrollment, treated with high-dose trivalent inactivated influenza vaccine (Fluzone HD) 2006-2007 formulation, Lot 3
- Active Comparator (Standard Fluzone®): Participants aged 65 years or older at enrollment, treated with standard Fluzone® vaccine 2006-2007 formulation
Period: Overall Study
Arm/Group | High-Dose Inactivated, Split-Virion Influenza Vaccine Lot 1 | High-Dose Inactivated, Split-Virion Influenza Vaccine Lot 2 | High-Dose Inactivated, Split-Virion Influenza Vaccine Lot 3 | Active Comparator (Standard Fluzone®)
Started | 857 | 848 | 870 | 1262
Completed | 848 | 847 | 868 | 1252
Not Completed | 9 | 1 | 2 | 10
Not completed — Serious Adverse Events | 1 | 0 | 1 | 4
Not completed — Protocol Violation | 2 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 5
Not completed — Withdrawal by Subject | 5 | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | High-Dose Inactivated, Split-Virion Influenza Vaccine Lot 1 | High-Dose Inactivated, Split-Virion Influenza Vaccine Lot 2 | High-Dose Inactivated, Split-Virion Influenza Vaccine Lot 3 | Active Comparator (Standard Fluzone®) | Total
Number analyzed (Participants) | 855 | 848 | 870 | 1260 | 3833
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0
  >=65 years | 855 | 848 | 870 | 1260 | 3833
Age, Continuous [Mean (Standard Deviation); unit: Years] | 72.9 (6.15) | 72.9 (6.20) | 72.9 (6.17) | 72.9 (5.99) | 72.9 (6.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 437 | 438 | 445 | 688 | 2008
  Male | 418 | 410 | 425 | 572 | 1825
Region of Enrollment [Number; unit: participants]
  United States | 855 | 848 | 870 | 1260 | 3833

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Titers (GMTs) of Hemagglutination Inhibition Antibody Titers Pre- and Post-vaccination With Fluzone® High Dose or Standard Fluzone® Vaccines.
Description: Antibodies against each of three Influenza antigens (virus) in Fluzone® High-Dose and Standard Fluzone® vaccines (A/H1N1 New-Caledonia; A/H3N2 Wisconsin; and B Malaysia) were determined by the Hemagglutination inhibition assay method.
Time Frame: Day 0 and Day 28 Post-vaccination
Population: The geometric mean titers was assessed in the Full Analysis Set according to the vaccine the subjects were randomized to receive. A total of 3851 participants were included in this analysis.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | High-Dose Inactivated, Split-Virion Influenza Vaccine Lot 1 | High-Dose Inactivated, Split-Virion Influenza Vaccine Lot 2 | High-Dose Inactivated, Split-Virion Influenza Vaccine Lot 3 | Active Comparator (Standard Fluzone®)
Number analyzed (Participants) | 854 | 861 | 861 | 1275
Titers
  A/H1N1 New Caledonia Pre-Dose | 28.25 [26.37 to 30.26] | 29.41 [27.39 to 31.57] | 27.86 [25.94 to 29.93] | 29.36 [27.72 to 31.11]
  A/H1N1 New Caledonia Post-Dose | 112.77 [105.64 to 120.37] | 114.63 [107.18 to 122.61] | 120.02 [112.12 to 128.48] | 67.29 [63.65 to 71.13]
  A/H3N2 Wisconsin Pre-Dose | 74.53 [67.29 to 82.55] | 77.3 [69.5 to 85.97] | 72.07 [65.12 to 79.77] | 74.74 [68.64 to 81.37]
  A/H3N2 Wisconsin Post-Dose | 595.03 [552.8 to 640.49] | 628.54 [583.21 to 677.4] | 603.59 [561.33 to 649.03] | 332.46 [310.44 to 356.05]
  B/Malaysia Pre-Dose | 19.24 [17.98 to 20.58] | 18.96 [17.71 to 20.29] | 19.78 [18.49 to 21.16] | 18.96 [17.93 to 20.04]
  B/Malaysia Post-Dose | 68.98 [64.77 to 73.47] | 69.26 [64.99 to 73.81] | 68.93 [64.81 to 73.3] | 52.34 [49.48 to 55.35]

2. Primary Outcome: Percentage of Participants With Seroconversion Post-vaccination With Fluzone® High-Dose or Standard Fluzone® Vaccines.
Description: Seroconversion was defined as a Hemagglutination Inhibition Antibody Titers of Titer ≥40 (1/dil) on Day 28 if pre-vaccination (Day 0) titer <10 (1/dil); or a four-fold increase of titer on Day 28, if pre-vaccination (Day 0) titer is ≥10 (1/dil) for each of the three Influenza vaccine antigens (A/H1N1 New-Caledonia; A/H3N2 Wisconsin; and B Malaysia).
Time Frame: Day 28 Post-vaccination
Population: The immunogenicity analysis was performed on the Full Analysis Set according to the vaccine the subjects were randomized to receive. A total of 3851 participants were included in this analysis.
Measure: Number; unit: Percentage of Participants
Arm/Group | High-Dose Inactivated, Split-Virion Influenza Vaccine Lot 1 | High-Dose Inactivated, Split-Virion Influenza Vaccine Lot 2 | High-Dose Inactivated, Split-Virion Influenza Vaccine Lot 3 | Active Comparator (Standard Fluzone®)
Number analyzed (Participants) | 854 | 861 | 861 | 1275
Percentage of Participants
  A/H1N1 New Caledonia | 47 | 47 | 52 | 23
  A/H3N2 Wisconsin | 70 | 68 | 70 | 51
  B/Malaysia | 43 | 41 | 42 | 30

3. Secondary Outcome: Percentage of Participants With Seroprotection Pre- and Post-Vaccination With Fluzone® High-Dose or Standard Fluzone® Vaccines.
Description: Seroprotection was defined as a Hemagglutination Inhibition Titers of at least 40 (≥ 1:40) for each of the Influenza vaccine antigens (A/H1N1 New-Caledonia; A/H3N2 Wisconsin; and B Malaysia) pre- or post-vaccination with Fluzone® High-Dose or Standard Fluzone® vaccines.
Time Frame: Day 0 and Day 28 Post-vaccination
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | High-Dose Inactivated, Split-Virion Influenza Vaccine Lot 1 | High-Dose Inactivated, Split-Virion Influenza Vaccine Lot 2 | High-Dose Inactivated, Split-Virion Influenza Vaccine Lot 3 | Active Comparator (Standard Fluzone®)
Number analyzed (Participants) | 854 | 861 | 861 | 1275
Percentage of Participants
  A/H1N1 New Caledonia Pre-Dose | 44 | 46 | 42 | 46
  A/H1N1 New Caledonia Post-Dose | 91 | 89 | 90 | 77
  A/H3N2 Wisconsin Pre-Dose | 70 | 69 | 68 | 69
  A/H3N2 Wisconsin Post-Dose | 99 | 99 | 99 | 97
  B/Malaysia Pre-Dose | 27 | 28 | 30 | 27
  B/Malaysia Post-Dose | 80 | 78 | 80 | 68

4. Secondary Outcome: Percentage of Participants Reporting Solicited Injection Site and Systemic Reactions After Fluzone® High-Dose or Standard Fluzone® Vaccination
Description: The occurrence, time to onset, number of days of occurrence, and severity of solicited injection site reactions: Injection Site Pain, Erythema, and Swelling; Solicited systemic reactions: Fever (temperature), Headache, Malaise, and Myalgia were collected.
Time Frame: Day 0 to Day 7 Post-vaccination
Population: The safety analysis was performed on the Full Analysis Set according to the participants who actually received a vaccine, whether or not the subject received the assigned vaccine. A total of 3,833 participants were included in the analysis set for the evaluation of all safety.
Measure: Number; unit: Percentage of Participants
Arm/Group | High-Dose Inactivated, Split-Virion Influenza Vaccine Lot 1 | High-Dose Inactivated, Split-Virion Influenza Vaccine Lot 2 | High-Dose Inactivated, Split-Virion Influenza Vaccine Lot 3 | Active Comparator (Standard Fluzone®)
Number analyzed (Participants) | 855 | 848 | 870 | 1260
Percentage of Participants
  Any Solicited Injection Site Reaction | 41 | 42 | 43 | 31
  Any Swelling | 9 | 9 | 9 | 6
  Grade 3 Swelling (≥ 5 cm) | 1 | 2 | 1 | 1
  Any Erythema | 16 | 15 | 14 | 11
  Grade 3 Erythema (≥ 5 cm) | 3 | 1 | 2 | 1
  Any Pain | 35 | 34 | 38 | 24
  Grade 3 Pain (Incapacitating) | 1 | 0 | 0 | 0
  Any Solicited Systemic Reaction | 37 | 33 | 33 | 29
  Any Fever | 4 | 3 | 4 | 2
  Grade 3 Fever (>102.2 ºF or >39.0 ºC) | 0 | 0 | 0 | 0
  Any Headache | 17 | 16 | 17 | 14
  Grade 3 Headache (Prevents Daily Activities) | 1 | 2 | 1 | 0
  Any Malaise | 20 | 18 | 16 | 14
  Grade 3 Malaise (Prevents Daily Activities) | 1 | 2 | 2 | 1
  Any Myalgia | 23 | 21 | 21 | 18
  Grade 3 Myalgia (Prevents Daily Activities) | 1 | 1 | 2 | 0

ADVERSE EVENTS:
Time Frame: Adverse events data were collected from day of vaccination (Day 0) for 6 months post-vaccination
Arm/Group | High-Dose Inactivated, Split-Virion Influenza Vaccine Lot 1 | High-Dose Inactivated, Split-Virion Influenza Vaccine Lot 2 | High-Dose Inactivated, Split-Virion Influenza Vaccine Lot 3 | Standad Dose Inactivated, Split-Virion Influenza Vaccine
Serious Adverse Events (participants affected / at risk) | 56/855 | 56/848 | 44/870 | 93/1260
Other Adverse Events (participants affected / at risk) | 455/855 | 454/848 | 449/870 | 544/1260
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High-Dose Inactivated, Split-Virion Influenza Vaccine Lot 1 (N=855) | High-Dose Inactivated, Split-Virion Influenza Vaccine Lot 2 (N=848) | High-Dose Inactivated, Split-Virion Influenza Vaccine Lot 3 (N=870) | Standad Dose Inactivated, Split-Virion Influenza Vaccine (N=1260)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Angina unstable (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 2 (2) | 1 (1) | 3 (3)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Cardiac Failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 4 (5) | 3 (3) | 0 (0) | 2 (2)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Congestive cardiomyopathy (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 2 (2) | 3 (3) | 0 (0) | 4 (4)
Coronary artery occlusion (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 2 (2) | 1 (1) | 2 (2) | 4 (4)
Ventricular fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrial septal defect (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal mass (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Crohn's disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Duodenitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Enterovesical fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 3 (3) | 1 (1)
Small intestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 2 (2) | 0 (0) | 5 (5)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hernia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Malaise (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Cholecystitis acute (Hepatobiliary disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chronic hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Cellulitis of male external genital organ (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 2 (2)
Extradural abscess (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 3 (3) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Implant site cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 6 (6) | 5 (6) | 6 (8) | 4 (4)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Staphylococcal infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Acetabulum fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back injury (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Device failure (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Head Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pacemaker complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Patella fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Perirenal haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Postoperative ileus (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Helicobacter pylori identification test positive (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gout (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Monarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (2)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Brain neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 2 (2) | 1 (1)
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchioloalveolar carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Non-hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oesophageal carcinoma (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Renal cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 5 (5) | 0 (0) | 1 (1)
Coordination abnormal (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Facial palsy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Grand mal convulsion (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Guillain-barre syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myasthenia gravis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Normal pressure hydrocephalus (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Parkinson's disease (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 5 (5)
Syncope vasovagal (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 1 (1) | 3 (4) | 4 (4)
Affective disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Bipolar I disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bipolar disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Drug dependence (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Renal failure chronic (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cystocele (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rectocele (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (4) | 0 (0) | 2 (2)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 3 (3) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aortic aneurysm (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral vascular disorder (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5.0% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High-Dose Inactivated, Split-Virion Influenza Vaccine Lot 1 (N=855) | High-Dose Inactivated, Split-Virion Influenza Vaccine Lot 2 (N=848) | High-Dose Inactivated, Split-Virion Influenza Vaccine Lot 3 (N=870) | Standad Dose Inactivated, Split-Virion Influenza Vaccine (N=1260)
Injection site erythema (General disorders) | 136 (136) | 125 (125) | 123 (123) | 136 (136)
Injection site pain (General disorders) | 295 (295) | 292 (292) | 328 (328) | 306 (306)
Injection site swelling (General disorders) | 79 (79) | 76 (76) | 75 (75) | 73 (73)
Malaise (General disorders) | 173 (173) | 150 (150) | 139 (139) | 176 (176)
Myalgia (Musculoskeletal and connective tissue disorders) | 197 (197) | 175 (175) | 178 (178) | 230 (230)
Headache (Nervous system disorders) | 146 (146) | 138 (138) | 147 (147) | 182 (182)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.